CLINICAL TRIAL: NCT03058536
Title: Progesterone and Cervical Pessary in Twins : A Prospective and Randomized Study to Prevent Preterm Birth (PRECEPT)
Brief Title: Progesterone and Cervical Pessary in Twins
Acronym: PRECEPET
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mario Henrique Burlacchini de Carvalho (Other)
Responsible Party: Sponsor-Investigator, Mario Henrique Burlacchini de Carvalho, Professor Doutor, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1.847.411
Record Dates: First submitted 2017-02-05; First posted 2017-02-23 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2017-02

CONDITIONS: Preterm Birth; Twin Pregnancy With Antenatal Problem
Keywords: twin short cervix pessary progesterone preterm birth
MeSH Terms: conditions — Premature Birth | interventions — Utrogestan; Progesterone

STUDY DESIGN:
Intervention Model Description: 312 twin pregnant women with short cervix between 16 and 27 weeks and 6 days of gestacional age will be randomized in four groups: daily 400mg vaginal progesterone combined with insertion of cervical pessary; isolated use of daily 400mg vaginal progesterone, isolated insertion of cervical pessary or expectant management (no intervention).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Progesterone (Active Comparator): 400 mg micronized vaginal progesterone daily from randomization to 36 weeks
  Interventions: Drug: Vaginal Progesterone
- Arabin Pessary and Progesterone (Active Comparator): Arabin Pessary and Natural Micronized Progesterone
  400 mg micronized vaginal progesterone daily from randomization to 36 weeks
  The device will be placed at randomization and will be removed during the 36th week of gestacional (or earlier if indicated) in combination with vaginal progesterone.
  Interventions: Other: Arabin Pessary and Progesterone
- Arabin Pessary (Active Comparator): The device will be placed at randomization and will be removed during the 36th week of gestacional (or earlier if indicated) without vaginal progesterone use.
  Interventions: Device: Arabin Pessary
- No intervention (No Intervention): Expectant management

INTERVENTIONS:
Device: Arabin Pessary — The cervical pessary will be inserted at the randomization and removed during the 36 week of pregnancy, unless labour occurs sooner.
  Arms: Arabin Pessary
Drug: Vaginal Progesterone — Treatment with 400 mg micronized progesterone daily, until the day of randomization to 36 weeks of pregnancy.
  Other Names: Utrogestan
  Arms: Progesterone
Other: Arabin Pessary and Progesterone — Arabin Pessary and Progesterone The cervical pessary will be inserted at the randomization and removed during the 36 week of pregnancy, unless labour occurs sooner. Treatment with 400 mg Micronized progesterone daily, until the day of randomization to 36 weeks of pregnancy.
  Arms: Arabin Pessary and Progesterone

SUMMARY:
The aim of this randomized control trial is to determine wheter cervical pessary plus vaginal progesterone (400mg) reduce preterm birth less than 34 weeks of gestacion and improve perinatal outcome, among women presenting asyntomatic short cervix, in twin pregnancy.

DETAILED DESCRIPTION:
The frequency of twin pregnancies has increased significantly, especially because of the assisted reproduction and advanced maternal age at conception. The twin pregnancies are responsible for 25 % of all preterm birth. Consequently, twin pregnancies are more associated with perinatal mortality and morbidity when compared to single pregnancies. Additionally, the short cervix (< 25 mm) in singleton and twin pregnancies are associated with significantly increased preterm birth.

Randomized controlled trials in singleton pregnancies reported that profilatic cervical cerclage and vaginal progesterone reduce significantly the rate of early preterm birth. In twin pregnancies, vaginal progesterone and profilatic cerclage have been shown to be ineffective in prevention of preterm birth.

However, two individual pacient data meta-analyses reported in a subgroup of women with twin pregancies and short cervix, that vaginal progesterone reduce significantly adverse neonatal outcomes. Nowadays, the effet of cervical pessary is contraditory, mainly in women with short cervix.

This is a randomized prospective trial at São Paulo University Medical School. This trial will involve 312 women with twins pregnancies and short cervix between 16 and 27 weeks and 6 days of gestacional age. Women with twin pregnancy and short cervix ( defined according to the gestacional age ) will be assigned randomly to daily vaginal progesterone (400mg) combined with insertion of cervical pessary, isolated use of daily vaginal progesterone (400mg) isolated insertion of cervical pessary or expectant management (no intervention). The primary outcome is to compare the rate of spontaneous delivery < 34 weeks of gestacion between groups.The secondary outcome is to compare the neonatal adverse outcome between the groups.

The aim of this study is to test the hypothesis that the insertion of a cervical pessary combined with vaginal progesterone, in twin pregnancies with short cervix would reduce the spontaneus preterm birth < 34 weeks' gestation.

ELIGIBILITY:
Inclusion Criteria:

* Twin pregnancy ( dichorionic or monochorionic diamniotic)
* Both fetuses alive
* Asymptomatic short cervix according to gestational age ( measurement less or equal 30 mm between 16 weeks + 0 day and 22 weeks + 0 day, less or equal 25 mm between 22 weeks + 1 day and 24 weeks + 0 day and less or equal 20 mm between 24 weeks + 1 day and 27 weeks + 6 days)
* Gestational age between 16 to 27weeks and 6 days
* Intact membranes
* Informed consent

Exclusion Criteria:

* Monoamniotic twins
* Twin Twin transfusion syndrome
* Rupture membranes
* Major malformation or chromosomal abnormality at least one fetus
* Women with Cervical cerclage in the current pregnancy
* Ballooning of membranes outside the cervix into the vagina
* Placenta previa
* Treatment with progesterone before randomization
* Allergy of the excipientes of the micronized progesterone
* Labor
* Severe hepatic disfunction, porphyria, otosclerosis, severe depression
* Use of drugs that interfere the effects of progesterone

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — pregnant women
Enrollment: 312 (Estimated)
Dates: Start 2017-02-21 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Preterm birth | 5 months
  Rate of preterm birth before 34 weeks gestation

SECONDARY OUTCOMES:
Neonatal Complications Rate | between birth and 28 days of age
  Includes necrotizing enterocolitis, intraventricular hemorrhage (grade 3 or higher), respiratory distress syndrome, retinopathy, sepsis, use of mechanical ventilation, time of hospitalization, and neonatal death.
Months from Randomization to delivery interval | 6 months
  Randomization may begin at 16 weeks, and most patient will be delivered between 36 and 38 weeks gestation.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Henrique Burlacchini de Carvalho, PhD, Principal Investigator — Hospital das Clínicas Universidade de São Paulo
Locations (1):
- Hospital das Clinicas da FMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kindinger LM, Poon LC, Cacciatore S, MacIntyre DA, Fox NS, Schuit E, Mol BW, Liem S, Lim AC, Serra V, Perales A, Hermans F, Darzi A, Bennett P, Nicolaides KH, Teoh TG. The effect of gestational age and cervical length measurements in the prediction of spontaneous preterm birth in twin pregnancies: an individual patient level meta-analysis. BJOG. 2016 May;123(6):877-84. doi: 10.1111/1471-0528.13575. Epub 2015 Sep 1. PMID 26333191
- [Background] Romero R, Nicolaides K, Conde-Agudelo A, Tabor A, O'Brien JM, Cetingoz E, Da Fonseca E, Creasy GW, Klein K, Rode L, Soma-Pillay P, Fusey S, Cam C, Alfirevic Z, Hassan SS. Vaginal progesterone in women with an asymptomatic sonographic short cervix in the midtrimester decreases preterm delivery and neonatal morbidity: a systematic review and metaanalysis of individual patient data. Am J Obstet Gynecol. 2012 Feb;206(2):124.e1-19. doi: 10.1016/j.ajog.2011.12.003. Epub 2011 Dec 11. PMID 22284156
- [Background] Norman JE, Mackenzie F, Owen P, Mactier H, Hanretty K, Cooper S, Calder A, Mires G, Danielian P, Sturgiss S, MacLennan G, Tydeman G, Thornton S, Martin B, Thornton JG, Neilson JP, Norrie J. Progesterone for the prevention of preterm birth in twin pregnancy (STOPPIT): a randomised, double-blind, placebo-controlled study and meta-analysis. Lancet. 2009 Jun 13;373(9680):2034-40. doi: 10.1016/S0140-6736(09)60947-8. PMID 19523680
- [Background] Brizot ML, Hernandez W, Liao AW, Bittar RE, Francisco RPV, Krebs VLJ, Zugaib M. Vaginal progesterone for the prevention of preterm birth in twin gestations: a randomized placebo-controlled double-blind study. Am J Obstet Gynecol. 2015 Jul;213(1):82.e1-82.e9. doi: 10.1016/j.ajog.2015.02.021. Epub 2015 Feb 27. PMID 25731690
- [Background] Schuit E, Stock S, Rode L, Rouse DJ, Lim AC, Norman JE, Nassar AH, Serra V, Combs CA, Vayssiere C, Aboulghar MM, Wood S, Cetingoz E, Briery CM, Fonseca EB, Worda K, Tabor A, Thom EA, Caritis SN, Awwad J, Usta IM, Perales A, Meseguer J, Maurel K, Garite T, Aboulghar MA, Amin YM, Ross S, Cam C, Karateke A, Morrison JC, Magann EF, Nicolaides KH, Zuithoff NP, Groenwold RH, Moons KG, Kwee A, Mol BW; Global Obstetrics Network (GONet) collaboration. Effectiveness of progestogens to improve perinatal outcome in twin pregnancies: an individual participant data meta-analysis. BJOG. 2015 Jan;122(1):27-37. doi: 10.1111/1471-0528.13032. Epub 2014 Aug 22. PMID 25145491
- [Background] Rode L, Klein K, Nicolaides KH, Krampl-Bettelheim E, Tabor A; PREDICT Group. Prevention of preterm delivery in twin gestations (PREDICT): a multicenter, randomized, placebo-controlled trial on the effect of vaginal micronized progesterone. Ultrasound Obstet Gynecol. 2011 Sep;38(3):272-80. doi: 10.1002/uog.9093. PMID 21739497
- [Background] Goya M, de la Calle M, Pratcorona L, Merced C, Rodo C, Munoz B, Juan M, Serrano A, Llurba E, Higueras T, Carreras E, Cabero L; PECEP-Twins Trial Group. Cervical pessary to prevent preterm birth in women with twin gestation and sonographic short cervix: a multicenter randomized controlled trial (PECEP-Twins). Am J Obstet Gynecol. 2016 Feb;214(2):145-152. doi: 10.1016/j.ajog.2015.11.012. Epub 2015 Nov 25. PMID 26627728
- [Background] Liem S, Schuit E, Hegeman M, Bais J, de Boer K, Bloemenkamp K, Brons J, Duvekot H, Bijvank BN, Franssen M, Gaugler I, de Graaf I, Oudijk M, Papatsonis D, Pernet P, Porath M, Scheepers L, Sikkema M, Sporken J, Visser H, van Wijngaarden W, Woiski M, van Pampus M, Mol BW, Bekedam D. Cervical pessaries for prevention of preterm birth in women with a multiple pregnancy (ProTWIN): a multicentre, open-label randomised controlled trial. Lancet. 2013 Oct 19;382(9901):1341-9. doi: 10.1016/S0140-6736(13)61408-7. Epub 2013 Aug 5. PMID 23924878
- [Background] Fox NS, Gupta S, Lam-Rachlin J, Rebarber A, Klauser CK, Saltzman DH. Cervical Pessary and Vaginal Progesterone in Twin Pregnancies With a Short Cervix. Obstet Gynecol. 2016 Apr;127(4):625-630. doi: 10.1097/AOG.0000000000001300. PMID 26959202
- [Background] Nicolaides KH, Syngelaki A, Poon LC, de Paco Matallana C, Plasencia W, Molina FS, Picciarelli G, Tul N, Celik E, Lau TK, Conturso R. Cervical pessary placement for prevention of preterm birth in unselected twin pregnancies: a randomized controlled trial. Am J Obstet Gynecol. 2016 Jan;214(1):3.e1-9. doi: 10.1016/j.ajog.2015.08.051. Epub 2015 Aug 28. PMID 26321037